CLINICAL TRIAL: NCT03448939
Title: A Phase 3 Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study of S5G4T-1 in the Treatment of Papulopustular Rosacea
Brief Title: A Study of S5G4T-1 in the Treatment of Papulopustular Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGT-54-01
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Papulopustular Rosacea
Keywords: papulopustular rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S5G4T-1 (Experimental): Participants will topically apply S5G4T-1 cream, once daily to face for 12 weeks.
  Interventions: Drug: S5G4T-1
- S5G4T-2 Vehicle Cream (Placebo Comparator): Participants will topically apply S5G4T-2 vehicle cream, once daily to face for 12 weeks.
  Interventions: Drug: S5G4T-2

INTERVENTIONS:
Drug: S5G4T-1 — Once a day topical cream
  Other Names: Encapsulated benzoyl peroxide (E-BPO) cream
  Arms: S5G4T-1
Drug: S5G4T-2 — Once a day topical cream
  Other Names: Vehicle cream
  Arms: S5G4T-2 Vehicle Cream

SUMMARY:
To assess the efficacy and safety of S5G4T-1 compared to its vehicle when applied once daily for 12 weeks in participants with papulopustular rosacea.

DETAILED DESCRIPTION:
In this Phase 3, double-blind, vehicle-controlled, parallel-group pivotal study, participants will be admitted only after a written informed consent has been obtained and after all inclusion/exclusion criteria have been met. Male and female participants at least 18 years of age with moderate or severe papulopustular rosacea will be eligible for enrollment for daily treatment with S5G4T-1 or its vehicle for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign an Institutional Review Board (IRB) approved written informed consent for this study.
2. Male and female 18 years of age and older.
3. Participants must have clinical diagnosis of moderate to severe rosacea.
4. Have a minimum total of 15 and a maximum of 70 total inflammatory lesions (papules and/or pustules) including those present on the nose.
5. Have 2 nodules or less.

Exclusion Criteria:

1. Females, who are pregnant, breastfeeding, or planning a pregnancy within the period of their study participation or were found to have positive pregnancy test at Baseline or screening visits.
2. Presence of more than 2 facial nodules or any nodule greater than 1 centimeter (cm).
3. Current or past ocular rosacea (for example, conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sol-Gel, Tampa, Florida, United States

REFERENCES:
- [Derived] Bhatia ND, Werschler WP, Baldwin H, Sugarman J, Green LJ, Levy-Hacham O, Nov O, Ram V, Stein Gold L. Efficacy and Safety of Microencapsulated Benzoyl Peroxide Cream, 5%, in Rosacea: Results From Two Phase III, Randomized, Vehicle-Controlled Trials. J Clin Aesthet Dermatol. 2023 Aug;16(8):34-40. PMID 37636253

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either S5G4T-1 (Encapsulated Benzoyl Peroxide [E-BPO] cream) or vehicle in a 2:1 ratio.
Groups:
- S5G4T-1: Participants topically applied S5G4T-1 cream, once daily to face for 12 weeks.
- S5G4T-2 Vehicle Cream: Participants topically applied S5G4T-2 vehicle cream, once daily to face for 12 weeks.
Period: Overall Study
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream
Started | 243 | 118
Received at Least 1 Dose of Study Drug | 239 | 113
Completed | 222 | 107
Not Completed | 21 | 11
Not completed — Adverse Event | 5 | 1
Not completed — Lost to Follow-up | 6 | 6
Not completed — Pregnancy | 1 | 1
Not completed — Withdrawal by Subject | 9 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all randomized participants who were dispensed study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream | Total
Number analyzed (Participants) | 243 | 118 | 361
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (13.21) | 52.4 (13.26) | 52.7 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 83 | 266
  Male | 60 | 35 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 39 | 125
  Not Hispanic or Latino | 156 | 77 | 233
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 233 | 116 | 349
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Baseline Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesions] — Inflammatory lesions were characterized as papules and pustules. A papule was defined as a solid, elevated inflammatory lesion equal to or less than 5 millimeter (mm) in diameter. A pustule was defined as an elevated inflammatory lesion equal to or less than 5 mm in diameter and contains pus (yellow-white exudate).
  lesions | 25.7 (11.07) | 26.3 (12.45) | 25.9 (11.52)
Baseline Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — Investigator's Global Assessment (IGA), where Investigator's rated the participant's acne from 0 (Clear) to 4 (Severe). A higher score indicated an increase in severity of facial acne.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 210 | 104 | 314
    4 - Severe | 33 | 14 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an IGA Score of Clear or Almost Clear From Baseline at Week 12
Description: Percentage of participants in each treatment group achieving an acne severity IGA score of "clear (score=0)" or "almost clear (score=1)".
Time Frame: Baseline through Week 12
Population: The ITT population consisted of all randomized participants who were dispensed study drug. Multiple imputation (Markov Chain Monte Carlo [MCMC]) was used to impute missing values.
Measure: Number; unit: Percentage of Participants
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream
Number analyzed (Participants) | 243 | 118
Percentage of Participants | 43.5 | 16.1

2. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts at Week 12
Description: Inflammatory lesions were characterized as papules and pustules. A papule was defined as a solid, elevated inflammatory lesion equal to or less than 5 mm in diameter. A pustule was defined as an elevated inflammatory lesion equal to or less than 5 mm in diameter and contains pus (yellow-white exudate). Least squares means and standard deviations from an analysis of covariance (ANCOVA) with factors of treatment, analysis center and treatment by analysis center interaction and the Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.
Time Frame: Baseline, Week 12
Population: The ITT population consisted of all randomized participants who were dispensed study drug. MCMC was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream
Number analyzed (Participants) | 243 | 118
Inflammatory Lesions | -17.4 (9.30) | -9.5 (9.45)

3. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream
Number analyzed (Participants) | 243 | 118
Percent Change | -68.2 (36.94) | -38.3 (37.02)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through end of study (Week 12)
Description: Safety population included randomized participants who were presumed to have used the study drug at least once and who provided at least 1 post-baseline safety evaluation.
Arm/Group | S5G4T-1 | S5G4T-2 Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/239 | 1/113
Other Adverse Events (participants affected / at risk) | 13/239 | 5/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S5G4T-1 (N=239) | S5G4T-2 Vehicle Cream (N=113)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S5G4T-1 (N=239) | S5G4T-2 Vehicle Cream (N=113)
Nasopharyngitis (Infections and infestations) | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Application site erythema (General disorders) | 8 | 2
Application site pain (General disorders) | 5 | 2
Application site pruritus (General disorders) | 3 | 1
Application site papules (General disorders) | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the Principal Investigator is not permitted to discuss or publish trial results without Sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03448939/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03448939/SAP_001.pdf